CLINICAL TRIAL: NCT00354601
Title: A Phase II Study of Weekly Docetaxel and Capecitabine for Persistent or Recurrent Platinum Resistant Epithelial Carcinoma of the Ovary, Fallopian Tube or Peritoneum
Brief Title: Docetaxel and Capecitabine in Treating Patients With Recurrent or Persistent Ovarian Epithelial Cancer, Fallopian Tube Cancer, or Peritoneal Cavity Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: funding withdrawn
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCCWFU-83203; CCCWFU-83203; CCCWFU-BG05-536; AVENTIS-CCCWFU-83203; CDR0000489036; ROCHE-CCCWFU-BG05-536
Record Dates: First submitted 2006-07-19; First posted 2006-07-20 (Estimated); Results first posted 2009-05-18 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-03

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Peritoneal Cavity Cancer
Keywords: fallopian tube cancer; peritoneal cavity cancer; recurrent ovarian epithelial cancer; ovarian clear cell cystadenocarcinoma; ovarian endometrioid adenocarcinoma; ovarian mucinous cystadenocarcinoma; ovarian serous cystadenocarcinoma; ovarian undifferentiated adenocarcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Capecitabine; Docetaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Weekly Docetaxel and Capecitabine (Experimental): Weekly Docetaxel and Capecitabine
  Interventions: Drug: capecitabine; Drug: docetaxel

INTERVENTIONS:
Drug: capecitabine — oral capecitabine twice daily on days 1-21
Drug: docetaxel — docetaxel IV over 30 minutes on days 1, 8, and 15

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving docetaxel together with carboplatin may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving docetaxel together with capecitabine works in treating patients with recurrent or persistent ovarian epithelial cancer, fallopian tube cancer, or peritoneal cavity cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate in patients with recurrent or persistent ovarian epithelial cancer, fallopian tube cancer, or peritoneal cavity cancer treated with docetaxel and capecitabine.

Secondary

* Determine the time to progression in patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.
* Determine the quality of life during treatment of these patients.

OUTLINE: Patients receive docetaxel IV over 30 minutes on days 1, 8, and 15 and oral capecitabine twice daily on days 1-21. Treatment repeats every 28 days for ≥ 6 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, on day 1 of each course, and then at completion of study treatment.

After completion of study treatment, patients are followed every 2-3 months.

ELIGIBILITY:
Inclusion Criteria:

DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Ovarian epithelial adenocarcinoma
  * Fallopian tube cancer
  * Peritoneal cavity cancer
* Recurrent or persistent disease after no more than 2 prior treatment regimens (1 regimen for primary disease and/or 1 regimen for recurrent disease)
* Platinum-resistant disease, defined as 1 of the following:

  * Treatment-free interval < 6 months after platinum-based therapy
  * Disease progression during platinum-based therapy
* Measurable disease by physical exam, chest x-ray, CT scan, or MRI
* No brain metastases

PATIENT CHARACTERISTICS:

* Gynecologic Oncology Group performance status 0-2
* Life expectancy > 6 months
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 8 g/dL
* Creatinine clearance ≥ 50 mL/min
* Bilirubin normal
* AST or ALT and alkaline phosphatase (AP) meeting 1 of the following criteria:

  * AST or ALT ≤ 5 times upper limit of normal (ULN) AND AP normal
  * AST or ALT ≤ 1.5 times ULN AND AP ≤ 2.5 times ULN
  * AST or ALT normal AND AP ≤ 5 times ULN
* No peripheral neuropathy > grade 2
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after completion of study treatment
* No other concurrent malignancy except for curatively treated nonmelanoma skin cancer
* No prior invasive malignancy < 5 years after curative therapy
* No serious uncontrolled medical or psychiatric illness that would preclude study participation or limit survival to < 6 months
* No history of severe hypersensitivity reaction to drugs formulated with polysorbate 80 or to fluoropyrimidine therapy or fluorouracil
* No inability to tolerate oral medication due to bowel obstruction, lack of physical integrity of the upper gastrointestinal tract, inability to swallow, or malabsorption syndrome
* No serious concurrent infections
* No clinically significant cardiac disease not well controlled with medication, including any of the following:

  * Congestive heart failure
  * Symptomatic coronary artery disease
  * Symptomatic cardiac arrhythmias
  * Myocardial infarction within the past 12 months

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior docetaxel or capecitabine or other fluoropyrimidine therapy
* Recovered from prior therapy
* At least 2 weeks since prior major surgery
* At least 4 weeks since prior chemotherapy, hormone therapy, or radiotherapy
* No other concurrent chemotherapeutic agents, biological therapy, radiotherapy, or other investigational agents

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2006-01; Primary Completion 2008-05 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte E. Miller, MD, Study Chair — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled 01/23/2006 to 03/16/2007 at which time the protocol was suspended for lack of funding
Groups:
- Docetaxel and Capecitabine: Docetaxel and Capecitabine therapy per protocol
Period: Overall Study
Arm/Group | Docetaxel and Capecitabine
Started | 2
Completed | 0
Not Completed | 2
Not completed — Protocol Violation | 1
Not completed — progression | 1

BASELINE CHARACTERISTICS:
Arm/Group | Docetaxel and Capecitabine
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.15 (8.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Secondary Outcome: Time to Progression
Description: Progression is defined as a 20% increase in tumor size of all the target lesions along the longest diameter
Time Frame: Evaluated every 8 weeks during treatment
Population: unable to analyze due to failure to complete treatment or study
Arm/Group | Docetaxel and Capecitabine
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Participants With Grade 3 or Higher Toxicity
Description: summary of grade 3 (per Common Toxicity Criteria) or higher toxicities which generally is described as a severe adverse reaction or symptom.
Time Frame: Days 1, 8, 15, 21 of each course and treatment end (28 days after last dose or start of new therapy)
Population: tracked during incomplete treatment period
Measure: Number; unit: participants
Arm/Group | Docetaxel and Capecitabine
Number analyzed (Participants) | 2
participants | 1

3. Secondary Outcome: Quality of Life
Description: comparison of treatment end to pre entry and day 1 of each treatment cycle.
Time Frame: Pre-entry, day 1, treatment end
Population: neither patient completed study
Arm/Group | Docetaxel and Capecitabine
Number analyzed (Participants) | 0

4. Primary Outcome: Objective Tumor Response
Description: The number of partial and complete responders among all evaluable patients as defined using Response Evaluation Criteria in Solid Tumors guidelines
Time Frame: 8 weeks
Population: unable to measure due to failure to complete
Arm/Group | Docetaxel and Capecitabine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Docetaxel and Capecitabine
Serious Adverse Events (participants affected / at risk) | 1
Other Adverse Events (participants affected / at risk) | 2
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Docetaxel and Capecitabine
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 1/2 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Docetaxel and Capecitabine
Diarrhea (Gastrointestinal disorders) | 2/2 (2)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 2/2 (2)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2/2 (2)

LIMITATIONS AND CAVEATS:
Early closure due to discontinuation of funding

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No